CLINICAL TRIAL: NCT03280693
Title: Relationships Among Body Mass Index, Body Balance and Bone Mineral Density
Brief Title: Relationships Among Body Mass Index, Body Balance and Bone Mineral Density in Postmenopausal Women
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Azza Mohammed, Principal invstigator, Cairo University
Other Study IDs: P.T.REC/012/00731
Record Dates: First submitted 2017-09-04; First posted 2017-09-12 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Osteoporosis; Fall Patients; Postmenopausal Disorder
Keywords: Body mass index,; Bone density; Balance; Postmenopause
MeSH Terms: conditions — Osteoporosis | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diagnostic test — Body balance was assessed using Berg Balance Scale (BBS), while BMD of the lumbar spine was measured by dual energy X-ray absorptiometry (DEXA) scan.

SUMMARY:
Body composition, bone mineral density (BMD), and body balance are important factors that threaten postural control. They act as vital elements in the vicious circle that leads to fracture occurrence in elderly population, particularly postmenopausal women.

DETAILED DESCRIPTION:
* The purpose of the current study was to evaluate the relationships among body mass index (BMI), body balance, and BMD (g/cm²) in postmenopausal women to be able to identify risk factors for fractures.
* Forty-eight postmenopausal women participated in this study. Body balance was assessed using Berg Balance Scale (BBS), while BMD of the lumbar spine was measured by dual energy X-ray absorptiometry (DEXA) scan.

The positive correlation between body balance and BMD in the current study can be explained that balance is controlled by sensory input, central processing, and neuromuscular responses. The sensory components consist of the vestibular, visual, and proprioceptive systems. An effective motor response requires an intact neuromuscular system and sufficient muscle strength to return the COG within the BOS when balance is disturbed. Postural balance in individuals with osteoporosis is significantly worse than in healthy individuals. Moreover, it was determined that balance scores in individuals with osteoporosis were 11% worse than scores of healthy individuals. Furthermore, exaggerated thoracic kyphotic curve is not only a disfiguring effect of osteoporosis but may also play a significant role in gait disorder, instability, and risk of falls.

In addition, back pain has a harmful impact on both balance and functional mobility in women with osteoporosis. Individuals with back pain may reduce their level of physical activity and, as a result, become weak in muscles required for balance and functional mobility. Impairment of the musculoskeletal and/or the neuromuscular system may negatively affect both balance and functional mobility.

In the same context, it was proved that women with decreased BMD and increased thoracic kyphosis presented greater body sway in the anterior/posterior direction on the force platform indicating more displacement of foot center of pressure (COP). They also confirmed that postmenopausal women with low BMD and increased thoracic kyphosis depend more on the hip strategy to maintain their postural control. This in turn probably causes more displacement of foot COP, thus causing greater body sway in all directions in comparison with the ankle strategy. it was also showed that women with loss of bone mass and increased thoracic kyphosis presented less foot COP displacement in the AP direction compared with the control group (with normal bone mass and normal thoracic curve.

The current study results also revealed that BMI was negatively correlated with both BMD and body balance in postmenopausal women. This can be illustrated that obese elderly women are often afraid of falls and sustaining fractures, so they prefer immobility and minimize their physical activity as much as possible. Because bone is formed when needed and resorbed when not needed as known as Wolff's law, BMD decreases and osteopenia/osteoporosis develops. Low BMD affect bone health as it leads to fragile weak bone and this in turn disturbs postural control and body balance. Additionally, obese women fail to control their center of gravity (COG) within base of support (BOS) disturbing their postural control and body balance, increasing risk of falls and making them more liable to fractures.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal women with ages range from 50 to 60 years

Exclusion Criteria:

* participation in sports
* vertebrobasillar insufficiency
* poor diet

Ages: 50 Years to 60 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — The study is based on investigating changes in the measured variables in postmenopausal women
Study Population: Forty-eight postmenopausal women participated in this study. Their mean values of age, body mass, height, and BMI were 53.5 ± 2.75 y, 89.08 ± 12.3 Kg, 159.67.8 ± 2.54 cm, and 34.89 ± 4.89 Kg/m², respectively. Body balance was assessed using Berg Balance Scale (BBS), while BMD of the lumbar spine was measured by dual energy X-ray absorptiometry (DEXA) scan.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
correlation between BMI and body balance | 7 months
  correlation analysis between BMI and body balance
correlation between BMI and BMD | 7 months
  correlation analysis between BMI and BMD

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu-Ambrose T, Eng J, Khan K., Carter ND, McKay HA. Older women with osteoporosis have increased postural sway and weaker quadriceps strength than counterparts with normal bone mass: overlooked determinants of fracture risk? J Gerontol A Biol Sci Med Sci. 2003. 58 (9): 862-6. Shumway-Cook A, Brauer S, Woollacott M. Predicting the probability for falls in community-dwelling older adults using the timed up and go test. Phys Ther. 2000. 80(9): 896-903. Sinaki M, Brey RH, Hughes CA, Larson DR, Kaufman KR. Balance disorder and increased risk of falls in osteoporosis and kyphosis: significance of kyphotic posture and muscle strength. Osteoporos Int. 2005.16 (8):1004-10. Liu-Ambrose T, Eng JJ, Khan KM, Mallinson A, Carter ND, McKay HA. The influence of back pain on balance and functional mobility in 65 to 75 year old women with osteoporosis. Osteoporosis Int. 2002. 13 (11): 868-73. Lynn SG, Sinaki M, Westerlind KC. Balance characteristics of person with osteoporosis. Arch Phys Med Rehabil. 1997. 78 (3): 273-6. Frost HD. Wolff's law and bone's structural adaptations to mechanical usage: an overview for clinicians. The angle Orthod. 1994. 64 (3): 175-80. Taes YE, Lapauw B, Vanbillemont G, Bogaert V, De Bac¬quer D, Zmierczak H, et al. Fat mass is negatively associat¬ed with cortical bone size in young healthy male siblings. J Clin Endocrinol Metab. 2009; 94 (7): 2325-31.